CLINICAL TRIAL: NCT02967107
Title: Cold Snare Polypectomy Versus Endoscopic Mucosal Resection for Colonic Sessile Serrated Polyps - A Randomised Controlled Trial
Brief Title: Cold Snare Polypectomy Versus Endoscopic Mucosal Resection for Colonic Sessile Serrated Polyps
Acronym: CSP-EMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Clinical Professor of Medicine and Director of Endoscopy, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREC/15/WMEAD/507
Record Dates: First submitted 2016-08-13; First posted 2016-11-17 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer; Adenoma
Keywords: adenoma; colorectal cancer; polypectomy; colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cold snare polypectomy (Active Comparator): Cold snare resection, if necessary, multi-piece to resect sessile serrated adenoma (SSA) 8-20mm
  Interventions: Procedure: Cold snare polypectomy
- Endoscopic mucosal resection (Active Comparator): Endoscopic mucosal resection (EMR), if necessary, multi-piece to resect sessile serrated adenoma (SSA) 8-20mm
  Interventions: Procedure: Endoscopic mucosal resection

INTERVENTIONS:
Procedure: Cold snare polypectomy — Use of a polypectomy snare closed over a polyp without electrocautery
  Other Names: CSP
  Arms: Cold snare polypectomy
Procedure: Endoscopic mucosal resection — Use of injected chromogelofusine solution to raise a lesion prior to snare resection with electrocautery
  Other Names: EMR
  Arms: Endoscopic mucosal resection

SUMMARY:
Comparing the efficacy of cold snare polypectomy with endoscopic mucosal resection

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer and it remains the second most commonly diagnosed malignancy in Australia. Colonoscopic polypectomy reduces the incidence and mortality from CRC by disrupting the adenoma-carcinoma sequence. Screening for CRC has proven to be effective in reducing mortality and morbidity from CRC and has become common practice. Interval cancers (development of a CRC within 6 to 60 months of a colonoscopy) occur in 6% of patients and estimations showed that up to 27% of these are due to incomplete adenoma resection.

The serrated neoplasia pathway accounts for 20- 30% of sporadic cancers. Serrated precursor lesions are thought to be a major contributor to the relative failure of colonoscopy in the prevention of proximal colorectal cancer (CRC) and to the 5- 7% of CRCs which occur in the period after complete colonoscopy and prior to surveillance, termed 'interval' cancer.

In addition to being difficult to detect, sessile serrated polyps (SSPs) are more likely to be incompletely resected than conventional adenomas. The CARE study demonstrated that 31% of SSPs had remnant tissue in the resection defect compared with 7.2% of conventional adenomas, and in lesions greater than 10 mm in size, residual tissue remained in 47.5%. SSPs may have indistinct margins, and smaller lesions may prove difficult to entrap with the snare because of their flat nature. SSPs also may contain dysplastic foci within the lesion, with an endoscopic appearance indistinguishable from conventional adenomas, and the surrounding serrated component may be overlooked and incompletely resected if this is not recognized.

The technique of colonoscopic polypectomy is continually evolving, leading to better outcomes with regard to polyp detection rate, complete resection rate (CRR) of polyps, patient comfort, safety and cost-efficacy. Although colonoscopy is considered the 'gold standard' for detecting and removing polyps, the technique is still imperfect. Questions about best practice for polypectomy remain, so optimizing the technique is expected to lead to better patient outcomes. The optimal treatment of SSPs should be effective, safe and inexpensive.

Such lesions can be removed by cold snare polypectomy or by endoscopic mucosal resection. Cold snare polypectomy (CSP) is now common practice and has proven to be a safe and effective technique for removal of any small polyps (<10 mm). Because of their physical characteristics, use of thin wire snares leads to a fast tissue transection and ability to remove SSP relatively swiftly. The size of snares suitable for SSP CSP is approximately 9 mm. Thus lesions greater than this size would need to be removed in more than one piece, introducing the possibility of incomplete resection. Endoscopic mucosal resection (EMR) is well established for laterally spreading colorectal lesions. It involves submucosal injection and diathermy assisted snare resection by piecemeal or en-bloc depending on polyp size. En bloc resection is possible for lesions up to 20 mm and facilitates histopathological evaluation. EMR is more time consuming than CSP and may be associated with diathermy related complications such as postpolypectomy bleeding, perforation and pain. The most efficient and safe method of removal of SSP has not been established.

ELIGIBILITY:
Inclusion Criteria:

* - Patients able to give informed consent to involvement in trial. For patients who do not speak English, an interpreter will be asked to translate the informed consent
* Patients referred to Westmead and Auburn Hospital Endoscopy Unit for a colonoscopy for all indications
* Age > 18 years
* At least one SSP 8-20 mm beyond the rectosigmoid junction without any endoscopic features of malignancy
* At least one SSP 8-20 mm beyond the rectosigmoid junction that according to the proceduralist, can be removed safely using either CSP or EMR

Exclusion Criteria:

* Current use of antiplatelets (excluding aspirin) or anticoagulants which have not appropriately been interrupted according to the guidelines [21]
* Known coagulopathy
* Pregnancy
* If any doubt about the morphology of the polyp, the patient will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with residual or recurrent adenoma as assessed at surveillance endoscopy | 4-6 months

SECONDARY OUTCOMES:
Number of participants with bleeding after the EMR procedure has finished as assessed by telephone interview at 2 weeks | 2 weeks
Number of participants with residual or recurrent adenoma as assessed at admission or telephone interview at 2 weeks | 2 weeks
Number of participants with pain after EMR as assessed by VAS score and telephone interview at 2 weeks | 2 weeks
  Pain after EMR

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided